CLINICAL TRIAL: NCT05832047
Title: Aggressive Hydration With Lactated Ringer's Solution Versus Plasma Solution for the Prevention of Post ERCP (Endoscopic Retrograde Cholangiopancreatography) Pancreatitis : Multicenter, Double Blind, Randomized Controlled Trial
Brief Title: Aggressive Hydration With Lactated Ringer's Solution Versus Plasma Solution for the Prevention of Post ERCP Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Do Hyun Park (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Sponsor-Investigator, Do Hyun Park, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DHP_ALPS study
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Disease
Keywords: ERCP; Endoscopic retrograde cholangiopancreatography; Pancreatitis
MeSH Terms: conditions — Pancreatic Diseases; Pancreatitis | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma solution (Experimental): Plasma solution (HK inno.N Corp., Seoul, Republic of Korea) is a balanced crystalloid solution that contains the same ingredients as Plasma-Lyte A (Baxter International, Deer field, Ill) .
  Preprocedure hydration begins 30-90 min before ERCP with an infusion rate of 10 mL/kg. All the ERCP procedures are performed under sedation with balanced propofol sedation (incremental dose of propofol in combination with fixed doses of fentanyl and midazolam), without general anaesthesia. The infusion rate during ERCP and 30-60 min after ERCP is 3 mL/kg/hour and 10 mL/kg, respectively (in the case of a 10 mL/kg injection after the procedure, the injection should be stopped at the point where it is necessary to move from the endoscopy room to the ward after the procedure, and the injection rate can be changed to 3 mL/kg/hour).
  Interventions: Drug: Plasma solution (4-hour aggressive hydration); Drug: 8-hour aggressive hydration
- Lactated Ringer's solution (Active Comparator): Preprocedure hydration begins 30-90 min before ERCP with an infusion rate of 10 mL/kg. All the ERCP procedures are performed under sedation with balanced propofol sedation (incremental dose of propofol in combination with fixed doses of fentanyl and midazolam), without general anaesthesia. The infusion rate during ERCP and 30-60 min after ERCP is 3 mL/kg/hour and 10 mL/kg, respectively (in the case of a 10 mL/kg injection after the procedure, the injection should be stopped at the point where it is necessary to move from the endoscopy room to the ward after the procedure, and the injection rate can be changed to 3 mL/kg/hour).
  Interventions: Drug: Lactated Ringer solution (4-hour aggressive hydration); Drug: 8-hour aggressive hydration

INTERVENTIONS:
Drug: Plasma solution (4-hour aggressive hydration) — Aggressive hydration : 10 mL/kg injection within 30~90min before procedure, 3 mL/kg/hr fluid injection during procedure, 10 mL/kg injection within 30~60min after procedure, fluid, injection at 3 mL/kg/hr for 4 hours.
  Other Names: Plasma solution-A Inj.
  Arms: Plasma solution
Drug: Lactated Ringer solution (4-hour aggressive hydration) — Aggressive hydration : 10 mL/kg injection within 30~90min before procedure, 3 mL/kg/hr fluid injection during procedure, 10 mL/kg injection within 30~60min after procedure, fluid, injection at 3 mL/kg/hr for 4 hours.
  Other Names: Hartmann Solution inno.N
  Arms: Lactated Ringer's solution
Drug: 8-hour aggressive hydration — If patients experienced postprocedural abdominal pain Numerical Rating Scale (NRS score>3) or a worsening of abdominal pain compared with the pain before ERCP, the administration of study fluid continues until 8 hours (3 mL/kg/hr ) regardless of the results of serum amylase/lipase within 4 hours after ERCP because serum amylase/lipase within 4 hours after ERCP may have a result approximately 1-2 hours (5 hours-6 hours after ERCP) after blood sampling
  Other Names: 8-h AH

SUMMARY:
In the existing Aggressive hydration comparison study related to the prevention of post-ERCP pancreatitis (PEP), research bias may occur due to the lack of blinding between fluids, so in this study, the investigators will conduct a multicenter randomized comparative study in which the comparative fluids are double-blinded to observe differences between fluids in the preventive effect of pancreatitis that occurs after ERCP (endoscopic retrograde cholangiopancreatography).

A total of 844 patients scheduled for ERCP will be enrolled in this clinical trial and randomly assigned to the lactated Ringer's solution or to the Plasma solution in a 1:1 ratio. Eligible patients will receive study drug or control drug for up to 24 hours before and after ERCP implementation.

In previous comparative studies related to PEP prevention, research bias may have been introduced because of insufficient blinding of the treatment strategies, as well as instances where the evaluating investigator did not perform blinding. We are therefore conducting a multicenter, randomized comparative study double-blinded as to the two types of fluid (lactated Ringer's solution or plasma solution), and in which the endoscopists, outcome assessors and patients are blinded to the randomization allocation.

DETAILED DESCRIPTION:
Post-ERCP pancreatitis (PEP), which occurs in 2% to 15% of all patients undergoing ERCP and is treated conservatively with fasting and sufficient fluid supply according to the standards of care for general acute pancreatitis, and most patients improve within a few days without major complications. However, high-risk patients are more susceptible to PEP with incidence rates between 15% and 42%, and severe pancreatitis can develop in 11.4% of PEP cases with a 3% mortality rate. Therefore, there are significant unmet needs for PEP patients.

In this trial, all patients will receive aggressive hydration involving fluids that are commercially available and widely administered. The trial aims to minimize potential risks and has established routine safety monitoring to protect the participants.

In real practice, it is crucial to consider not just the type of fluid utilized, but also the most effective fluid volume for preventing PEP, along with the optimal timing for administering the fluid. Given that a significant number of ERCPs are performed in outpatient settings in the USA and other countries, the current protocol allowing outpatients to occupy recovery areas for extended periods, such as 8 hours post-ERCP, seems challenging to implement in real clinical practice. These considerations highlight the necessity for a re-evaluation of existing guidelines. Therefore, the present reassessment aims, not only to optimize efficiency and patient flow in medical settings but also to evaluate the effectiveness of the protocol in preventing PEP considering practical duration of intravenous fluid infusion, such as 4 hours postprocedure.

ELIGIBILITY:
Inclusion Criteria:

Among patients with naive major duodenal papilla in patients, we will include those who are at average-to-high risk of PEP (if one or more of the following criteria) after ERCP and agree to enroll in this clinical trial.

1. 40 years of age or younger
2. (Suspected) Sphincter of oddi dysfunction
3. The normal level of serum total bilirubin
4. History of recurrent pancreatitis
5. Require injection of a contrast agent into the pancreatic duct
6. Require endoscopic biliary or pancreatic sphincterotomy
7. Require precut sphincterotomy
8. Require endoscopic papillary balloon dilation
9. Planned endoscopic papillectomy
10. Diagnosed with periampullary tumor and planned for insertion of a self-expanding metal stent

Exclusion Criteria:

Subjects are excluded if they meet any of the following items.

1. Not consented to study participation
2. 18 years of age or younger
3. Severe comorbidities (e.g., end-stage kidney disease, end-stage chronic obstructive pulmonary disease, hypoglycemic dysregulation, decompensated cirrhosis)
4. Sepsis (defined as meeting two or more of the following items):

   * Body temperature >38.3ºC or <36ºC
   * Heart rate >90 beats/min
   * Tachypnea (respiratory rate > 20 breaths/min)
   * Leukocytosis (WBC>12,000/uL) or leukopenia (WBC<4000/uL)
5. Acute pancreatitis
6. Chronic pancreatitis
7. Heart failure (NYHA class 2 or higher)
8. Clinical signs of fluid overload
9. Hypernatremia (>150 mEq/L) or hyponatremia (<130 mEq/L)
10. History of endoscopic sphincterotomy
11. History of endoscopic papillary (balloon) dilation
12. Hypercalcemia or alkalemia
13. Scheduled for regular endoscopic biliary stent change
14. Patients with pancreatic head tumors and a presumed low risk for pancreatitis
15. Lack of access to the major duodenal papilla due to surgically altered anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of pancreatitis after ERCP | the next morning or within 24 hours after ERCP
  The new onset or worsening of pain in the upper abdomen, accompanied by an elevation of pancreatic enzymes to at least three times the upper normal level within 24 hours after the procedure, requiring hospitalization for a minimum of two nights.

SECONDARY OUTCOMES:
Occurrence of pancreatitis after ERCP at 4 hours after ERCP | 4 hours after ERCP
  The new onset or worsening of pain in the upper abdomen and the level of pancreatic enzymes is elevated>3 times the upper limit of normal level after 4 hours after ERCP
Number of Participants with Clinical signs of fluid overload | 4 hours and, and the next morning or within 24 hours after ERCP
  Clinical signs of fluid overload, for example, peripheral edema, pulmonary rales, increased jugular venous pressure, hepatojugular reflux, or both wll be monitored by investigator. If these signs are observed, hemodynamic testing or imaging studies will be done to investigate the evidence of pulmonary oedema, peripheral oedema, cardiac insufficiency and hypernatraemia.
Number of Participants with Asymptomatic Hyperamylasemia | 4 hours and, the next morning or within 24 hours after ERCP
  Elevated level of serum amylase without upper abdominal pain
Occurrence or aggravation of upper abdominal pain | 4 hours and, the next morning or within 24 hours after ERCP
  Occurrence or aggravation of upper abdominal pain
Days of ERCP-related hospital stay | Time for upper abdominal pain to disappear after the date of ERCP - up to 20 days
  Time for upper abdominal pain to disappear after the date of ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Seoul Hopital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho IR, Choi JH, Park JK, Huh G, Lee SH, Paik WH, Park DH. Aggressive hydration with lactated Ringer's solution versus plasma solution for the prevention of post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (ALPS study): protocol for a multicentre, double-blind, randomised controlled trial. BMJ Open. 2024 Jul 1;14(7):e084052. doi: 10.1136/bmjopen-2024-084052. PMID 38955368